CLINICAL TRIAL: NCT06066723
Title: A Cross-sectional Pilot Study of 19F MRI in Healthy Children and Children With Mild Cystic Fibrosis Lung Disease
Brief Title: 19F MRI in Healthy Children and Children With Mild Cystic Fibrosis Lung Disease
Status: Recruiting | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Cystic Fibrosis Foundation (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 23-0700; 5K23HL138257-03 (NIH)
Record Dates: First submitted 2023-09-20; First posted 2023-10-04 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-02

CONDITIONS: Cystic Fibrosis in Children
Keywords: 19F MRI; ventilation; pediatrics
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Children with CF: All subjects to receive inhaled perfluoropropane during MRI procedures, including standard breath hold and free-breathing technique. Subjects will breathe the gas for 5 breath hold cycles (variable volumes as lung capacity/size varies per participant).
  Interventions: Combination Product: 19F MRI
- Healthy Children: All subjects to receive inhaled perfluoropropane during MRI procedures, including standard breath hold and free-breathing technique. Subjects will breathe the gas for 5 breath hold cycles (variable volumes as lung capacity/size varies per participant).
  Interventions: Combination Product: 19F MRI

INTERVENTIONS:
Combination Product: 19F MRI — Inhalation of a biologically inert contrast gas, perfluoropropane, combined with 19F-tuned MRI with image acquisition at breath-hold and during tidal breathing.
  Other Names: PFP

SUMMARY:
This study capitalizes on the emerging technology of 19F MRI, using conventional 'thermally' polarized perfluorinated gas (perfluoropropane, or PFP) mixed with oxygen and studied with magnetic resonance imaging (MRI) to visualize ventilation. This technique has not been studied in children.

Children and adolescents (6-17 years old) with cystic fibrosis (CF) who have normal spirometry will undergo 19F MRI with the inhalation of an inert contrast gas to study ventilation. Comparisons will be made to a cohort of healthy children (6-17 years old) who will perform the same measures. The primary outcome measure is the feasibility of conducting these studies in the pediatric population. Parallel performance of multiple breath nitrogen washout (MBW) and spirometry will be used to compare the sensitivity of these outcomes to the presence of mild lung disease in these children. Finally, the investigators will compare data obtained during standard breath holds with a novel "free-breathing" technique that will eliminate the need for breath holds during MRI acquisition.

ELIGIBILITY:
Inclusion Criteria:

* 6-17 years old
* Non-smoker and non-vaper
* Cystic Fibrosis (CF) Group: must have a diagnosis of CF
* No use of supplemental oxygen
* They must be able to perform spirometry and have stable lung function (within 10% personal best in the last 6 months) and no exacerbations within the past 4 weeks
* Baseline forced expiratory volume in 1 second (FEV1) >80% with ratio of the forced expiratory volume in the first one second to the forced vital capacity of the lung (FEV1:FVC) ratio >0.7

Exclusion Criteria:

* Healthy volunteers: with any history of chronic lung disease (i.e. asthma)
* Active or former smoker with less than 1 year of quitting
* Unable to undergo an MRI of the lungs and chest because of contraindications, including:

  * Injury to the eye involving a metallic object
  * Injury to the body involving a metallic object
  * Presence of an implanted drug infusion device that is not MRI safe
  * Bone growth of fusion simulator
  * Presence of cochlear, otologic, or ear implant
  * Shunt (spinal or intraventricular)
  * Any implant held in place by magnet
  * Claustrophobia
* Unable to tolerate the inhalation of the gas mixture
* Facial hair preventing a tight fit of the mask used in the study
* Pregnancy
* Changes in medication that may affect CF lung disease or lung function in the past 28 days, including experimental therapies

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy volunteers between the ages of 6-17 years old without known lung disease OR people with cystic fibrosis between the ages of 6-17 years
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2025-06-16 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Participation rate | through study completion, recruitment for 2 years
  The number of eligible participants approached for the study divided by the number who consent to participate.
Completion rate | through study completion, recruitment for 2 years
  The number of consented participants divided by the number of participants who complete each portion of the study.
Parental acceptability score | Day 1, assessed at single visit
  Acceptability questionnaire for guardian; 2 questions, each on a 10 point Likert scale
  * Implementation: qualitative description of barriers encountered
  * Practicality: % of participants completing the study with research quality data
Child acceptability score | Day 1, assessed at single visit
  Acceptability questionnaire for participant; 2 questions, each on a 10 point Likert scale
  * Implementation: qualitative description of barriers encountered
  * Practicality: % of participants completing the study with research quality data

SECONDARY OUTCOMES:
MRI defined ventilation defect parameters (VDP) in healthy participants | Day 1, assessed at single visit
  The 19F Volumetric interpolated breath-hold examination (VIBE) scans and proton nuclear magnetic resonance imaging (1H-MRI) will be saved as Digital Imaging and Communications in Medicine (DICOM) images and imported to Medical Image Merge (MIM) software. The percentage of lung with ventilation defects (VDP) after the 5th inspiratory cycle will be measured, using the 95th percentile of background noise on the last wash-in scan as the threshold value defining absence of ventilation. The investigators will assess ventilation defect parameters (VDP) scored in healthy participants (mean + SD)
MRI defined fraction of lung volume with slow gas washout time (FLVlongtau2) in healthy participants | Day 1, assessed at single visit
  The 19F Volumetric interpolated breath-hold examination (VIBE) scans and 1H-MRI will be saved as Digital Imaging and Communications in Medicine (DICOM) images and imported to Medical Image Merge (MIM) software. The fraction of the total lung volume with slow gas wash-out kinetics (FLV↑tau2) will be calculated for lung regions without an overlapping full ventilation defect. The investigators will assess FLVlongtau2 scored in healthy participants (mean + SD)
MRI defined VDP in participants with cystic fibrosis | Day 1, assessed at single visit
  The 19F VIBE scans and 1H-MRI will be saved as Digital Imaging and Communications in Medicine (DICOM) images and imported to Medical Image Merge (MIM) software. The percentage of lung with ventilation defects (VDP) after the 5th inspiratory cycle will be measured, using the 95th percentile of background noise on the last wash-in scan as the threshold value defining absence of ventilation. The investigators will assess ventilation defect parameters (VDP) scored in participants with cystic fibrosis (mean + SD)
MRI defined fraction of lung volume with slow gas washout time (FLVlongtau2) in participants with cystic fibrosis | Day 1, assessed at single visit
  The 19F Volumetric interpolated breath-hold examination (VIBE) scans and 1H-MRI will be saved as Digital Imaging and Communications in Medicine (DICOM) images and imported to Medical Image Merge (MIM) software. The fraction of the total lung volume with slow gas wash-out kinetics (FLV↑tau2) will be calculated for lung regions without an overlapping full ventilation defect. The investigators will assess FLVlongtau2 scored in participants with cystic fibrosis (mean + SD)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Goralski, MD, Principal Investigator — UNC Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No